CLINICAL TRIAL: NCT01071434
Title: Investigating the Feasibility of Using Real-time Cine-MRI for Treating Moving and Deforming Tumors
Brief Title: Feasibility of Using Real-time Cine-MRI for Treating Moving & Deforming Tumors
Status: Terminated | Type: Observational
Why Stopped: PI left
Sponsor: Stanford University (Other)
Collaborators: The American Association of Physicists in Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: VAR0042; SU-06112009-2702 (Other: Stanford University)
Record Dates: First submitted 2009-12-16; First posted 2010-02-19 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Pancreatic Cancer; Liver Cancer; Lung Cancer; Lung Cancer Non-Small Cell Cancer (NSCLC); Lung Cancer Small Cell Lung Cancer (SCLC); Hepatobiliary Cancers; Hepatobiliary Cancers Liver; Hepatobiliary Cancers Hepatocellular Carcinoma (Hepatoma); Hepatobiliary Cancers Gallbladder; Hepatobiliary Cancers Bile Duct
MeSH Terms: conditions — Pancreatic Neoplasms; Liver Neoplasms; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Carcinoma, Hepatocellular | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: MR Imaging

SUMMARY:
This study aims to investigate and optimize imaging sequences and parameters of rapid real-time MRI in order to obtain adequate guidance for accurately and precisely delivering radiation to moving abdominal and thoracic tumors.

DETAILED DESCRIPTION:
Accurate dose delivery remains one of the weakest aspects of radiotherapy, especially in the case of thoracic and abdominal tumors, where significant patient motion occurs during dose delivery (intrafraction motion). Such motion results in geometric and dosimetric uncertainties that compromise treatment quality. Effective management of intrafraction motion is therefore key to realizing the full potential of modern image-guided radiation therapy (IGRT). While external markers have been found to be well-correlated with internal anatomy within an imaging session, there is no guarantee that these correlations will continue to exist and be constant throughout the course of the therapy. In general, implanted, radio-opaque seeds have been found to be more reliable than external markers. However, implantation of fiducials, whether radio-opaque or electromagnetic, is necessarily invasive and carries with it the risk of associated complications - an issue that becomes especially important for cancer patients with weakened immune systems. Currently, MR imaging is the only modality that is non-invasive and provides high quality volumetric information for the whole body.

The "ideal" intrafraction motion management requires complete spatio-temporal knowledge of the irradiated anatomy. However, to date, there is no clinical method of directly visualizing the tumor volume during dose delivery. Most techniques rely on external or internal surrogate markers which often provide (usually non-volumetric) information of limited accuracy and reliability. In addition, internal markers impose significant "costs" on the patient in terms of interventional complications and increased imaging dose. In this work, we investigate the feasibility of using in-room, fast cine MR imaging as a non-invasive means to provide real-time, soft-tissue-based, volumetric image guidance for continuous monitoring of the target and surrounding anatomy. To date, there has been no systematic investigation of the imaging requirements of an integrated MRI+linac for the specific task of real-time radiotherapy guidance.

ELIGIBILITY:
Inclusion Criteria:3.1.1. Eligible disease(s)/stage(s) AJCC Stage I, II, III or IV lung, liver or pancreatic cancer of any histology to be treated using radiotherapy will be eligible for this study.

3.1.2. Allowable type and amount of prior therapy  Any types and amounts of prior therapy will be allowed for this study.

3.1.3. Age restriction and/or gender/ethnic restrictions Patients must be greater than or equal to 18 years of age. There are no gender or ethnic restrictions.

3.1.4. Life expectancy restrictions  None.

3.1.5. ECOG or Karnofsky Performance Status  Karnofsky performance status of 50 or greater

3.1.6. Requirements for organ and marrow function  None.

3.1.7. Ability to understand and the willingness to sign a written informed consent document.

3.1.8. Pain-free in supine position Exclusion Criteria:3.2.1 Children (age <18)

3.2.2 Metallic implants, embedded metallic objects, implanted biomedical devices e.g., cardiac pacemakers

3.2.3 Women who are pregnant or trying to get pregnant

3.2.4 Pain in supine position

3.2.5 Karnofsky performance status < 50

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible disease(s)/stage(s) AJCC Stage I, II, III or IV lung, liver or pancreatic cancer of any histology to be treated using radiotherapy will be eligible for this study.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2009-02; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
investigate and optimize imaging sequences and parameters of rapid real-time MRI in order to obtain adequate guidance for accurately and precisely delivering radiation to moving abdominal and thoracic tumors. | two hours

CONTACTS AND LOCATIONS:
Overall Officials: Amit Sawant, Principal Investigator — Stanford University; Paul J Keall, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States